CLINICAL TRIAL: NCT05776017
Title: A Phase 1b/2b Double Blind, Randomized, Controlled Study of the Safety, Immunogenicity, and Efficacy of Malaria Vaccine Candidate MSP3-CRM-Vac4All/ Alhydrogel® in Young Children in Mali
Brief Title: MSP3-CRM-Vac4All/ Alhydrogel® Vaccine
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vac4All (Industry)
Collaborators: Malaria Research and Training Center, Bamako, Mali (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V4ALL/MSP3/009
Record Dates: First submitted 2023-02-25; First posted 2023-03-20 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Malaria,Falciparum
Keywords: malaria; malaria vaccine; vaccine efficacy
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Aluminum Hydroxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Vaccine recipients and their parent(s)/guardian(s) as well as all investigators and study personnel responsible for the vaccination, evaluation of safety and immunogenicity endpoints will all be unaware to the exact treatment given to the participant. Randomization will be programmed into the eCRF, as subjects are confirmed to be eligible for enrollment and to be vaccinated. A password protected electronic randomized vaccination allocation list will be sent to the designated vaccine pharmacist. The investigator will send a request for vaccination to the pharmacy using the subject randomization number (which will be the subject unique ID number) assigned by the eCRF. For each child, eligibility will have to be counter checked and signed by a second person before allocation of study ID number.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Vaccine (Experimental): MSP3-CRM-Vac4All/ Alhydrogel®
  Interventions: Biological: MSP3-CRM-Vac4All/ Alhydrogel®
- Control Vaccine (Active Comparator): Anti-rabies vaccine
  Interventions: Biological: Anti-Rabies Vaccine

INTERVENTIONS:
Biological: MSP3-CRM-Vac4All/ Alhydrogel® — 30 microgram MSP3-CRM-Vac4All protein extemporaneously formulated with Alhydrogel® adjuvant
  Arms: Test Vaccine
Biological: Anti-Rabies Vaccine — Control vaccine
  Arms: Control Vaccine

SUMMARY:
Two-arm, randomized, double-blinded and controlled clinical trial to first assess the safety and tolerability of the vaccine in a Phase 1b trial and proceed to assess its efficacy against clinical malaria in young children living in highly seasonal malaria areas of Mali

DETAILED DESCRIPTION:
This study is designed to be executed in two steps to achieve the primary efficacy objective:

The first step is a Phase 1b safety study, involving injections in a small safety subgroup for each dose before age-de-escalation into the younger age group and then proceeding to the second step of dosing the corresponding injection in the larger Phase 2b efficacy cohort.

Vaccination of the Phase 2b cohort will require an acceptable reactogenicity data over the first week following the corresponding vaccination of the older and younger age groups in the Phase 1 subgroup. The study DSMB will be charged with this review and ensuring that vaccination proceeds only if the reactogenicity profile meet study "go" criteria (Table 1).

The objectives of each phase are:

Phase 1b: The primary objective is to assess the safety and tolerability of the vaccine for each injection. The secondary objective is to evaluate the immune response to the vaccine and safety for up to 12 months after the first dose.

Phase 2b: The primary objective is to assess the efficacy in young children* against clinical malaria** during one transmission season. The timeline for the primary analysis assessment is from 14 days to 6 months after Dose 3.

Should the primary analysis data demonstrate that the vaccine gives good efficacy, a boost vaccination will be programmed to be administered to willing subjects before the start of the subsequent transmission season. The study protocol will be amended with the precise details in this event.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 12-59 months years old
* Healthy by medical history, physical examination and laboratory investigation
* Signed/thumb printed informed Consent by guardian/parent
* Resident in the study area villages during the whole trial period

Exclusion Criteria:

* Symptoms, physical signs of disease that could interfere with the interpretation of the trial results or compromising the health of the participants
* Immunosuppressive therapy (steroids, immune modulators or immune suppressors) within 3 months prior recruitment. (For corticosteroids, this will mean prednisone, or equivalent, more or equal to 0.5 mg/kg/day. Inhaled and topical steroids are allowed.)
* Cannot be followed for any social, psychological or geographical reasons.
* Use of any investigational drug or vaccine other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use up to 30 days after the third dose.
* Suspected or known hypersensitivity to any of the vaccine components or to previous vaccine.
* Clinically significant laboratory abnormalities on screened blood samples.
* Planned administration of a vaccine not foreseen by the study protocol within 30 days before the first dose of vaccine. An exception, is the receipt of an childhood immunization program or licensed vaccine (measles, oral polio, Hib, meningococcal and combined diphtheria/pertussis/tetanus vaccines) which may be given before or after vaccination*.
* Evidence of chronic or active hepatitis B or C infection
* Presence of chronic illness that, in the judgment of the investigator, would interfere with the study outcomes or pose a threat to the participant's health.
* Administration of immunoglobulin and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period
* History of surgical splenectomy.
* Moderate or severe malnutrition at screening based on clinical judgement.

  o (Weight-for-age Z score of less than -3 or other clinical signs of malnutrition).
* Previous participation to a malaria vaccine trial
* Known history of HIV infection

Ages: 12 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 465 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Protective Efficacy against Clinical Malaria | The timeline for assessment will be from 14 days to 6 months after Dose 3.
  To assess the efficacy of 30 µg MSP3-CRM-Vac4All/Alhydrogel® vaccine in children ages 12-60 months old, against clinical malaria occurring over one transmission season.
  The primary efficacy outcome is clinical malaria, with the primary case definition of clinical malaria episodes defined as a febrile episode with an axillary temperature of ≥ 37.5ºC with P. falciparum parasitemia ≥5000/µL

SECONDARY OUTCOMES:
Efficacy- different definitions of malaria fever and parasite thresholds on microscopy | For 12 months after first vaccination
  To compare efficacy against clinical malaria for different case definitions using
  * Fever thresholds that are higher than 37.5ºC, such as 38.5ºC and 39.5ºC
  * History of fever instead of measured fever
  * Different parasitemia by microscopy thresholds [any parasitemia, 1000, 10,000 and 20,000/µL]
  Efficacy outcomes
  * clinical malaria episodes defined as a febrile episode with an axillary temperature of ≥ 38.5ºC with P. falciparum parasitemia ≥5000/µL or ≥ 39.5ºC with P. falciparum parasitemia ≥5000/µL or
  * clinical malaria episodes defined as history of fever with P. falciparum parasitemia of the following levels: any parasitemia, 1000, 10,000 and 20,000/µL clinical malaria episodes defined as a febrile episode with an axillary temperature of ≥ 38.5ºC with or ≥ 39.5ºC with P. falciparum parasitemia of the following levels: any parasitemia, 1000, 10,000 and 20,000/µL
Efficacy duration | For 12 months following the first vaccination
  To assess the efficacy of MSP3-CRM-Vac4All/Alhydrogel® in young children against clinical malaria occurring during the 12 months following dose 3.
Efficacy against first malaria episodes | From 14 days post 2nd or 3rd vaccination to 6 months following and up to the end of study follow-up (12 months after first vaccination
  To assess the efficacy of MSP3-CRM-Vac4All/Alhydrogel® in young children against first clinical malaria episodes occurring from over the 6 month period 14 days after 2nd and 3rd vaccination and up to the end of study follow-up (12 months after first vaccination).
  The efficacy outcome is first episode of clinical malaria, with the case definition of clinical malaria episodes defined as a febrile episode with an axillary temperature of ≥ 37.5ºC with P. falciparum parasitemia ≥5000/µL
Efficacy (conditional boost) | For the 6 months following boost vaccination
  To assess the efficacy of MSP3-CRM-Vac4All/Alhydrogel® in young children against clinical malaria occurring The efficacy outcome is clinical malaria, with the primary case definition of clinical malaria episodes defined as a febrile episode with an axillary temperature of ≥ 37.5ºC with P. falciparum parasitemia ≥5000/µL
Efficacy (conditional boost) | For the 12 months following boost vaccination
  To assess the efficacy of MSP3-CRM-Vac4All/Alhydrogel® in young children against clinical malaria occurring.
  The efficacy outcome is clinical malaria, with the primary case definition of clinical malaria episodes defined as a febrile episode with an axillary temperature of ≥ 37.5ºC with P. falciparum parasitemia ≥5000/µL
Number of adverse events | During the month following each vaccination, and 6 months and 12 months after first vaccination.
  To assess the safety and reactogenicity of 3 doses of 30 µg MSP3-CRM-Vac4All/Alhydrogel® given at D0, D28 and D56 in healthy young children
Number of adverse events for conditional boost vaccination | At one month, 6 month and 12 months following boost vaccination
  Safety and reactogenicity of boost vaccination doses of MSP3-CRM-Vac4All/Alhydrogel® in healthy young children
Immune response | From 14 days post last dose to up to a month after last dose, 6 months after last dose and 12 months after first dose
  To examine the duration of immune responses of a 3-dose regimen of during periods corresponding to that used for primary and other secondary efficacy endpoints as measured through a > 5-fold decrease of MSP3-specific serum IgG antibody titers after each vaccination in comparison to baseline levels (14 days post last dose)
Immune response | A month after dose 3
  To determine immunogenicity in terms of the proportion with titres either more than 3SD above the median for negative controls (positive) or at least 50% of the positive controls (strongly positive) after dose 3.
Parasite densities | From vaccination to up to 6 months after last dose and 12 months after first dose.
  To measure effect on parasitemia by comparing parasite densities in malaria episodes occurring in vaccinees compared to control

CONTACTS AND LOCATIONS:
Overall Officials: Manamadou Thera, MD, Study Director — MRTC, University of Sciences Techniques and Technologies of Bamako, Mali Locations:
Locations (1):
- Malaria Research and Training Center (MRTC), University of Sciences Techniques and Technologies of Bamako, Mali, Bamako, Mali

IPD SHARING:
Plan to Share IPD: No